CLINICAL TRIAL: NCT03482518
Title: Effectiveness of Postural Insoles Adapted in Slippers for People With Persistent Heel Pain and Metatarsalgias: a Clinical, Controlled, Randomized and Double Blind Study
Brief Title: Effectiveness of Postural Insoles Adapted in Slippers for People With Persistent Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, Assistant professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRNCHINELOS
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Heel Pain Syndrome; Metatarsalgia
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants will be informed that they will be drawn to participate in one of the two groups (intervention group or control group). Allocation in the groups will be done randomly, by lot, following the order of randomization, keeping the confidentiality, ie, one should not know to which group the participant will be sent before he / she agrees to be evaluated and sign the TCLE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group volunteers will receive a pair of custom slippers with perforated synthetic leather cover with elements in insoles. They will be advised to wear the slipper for 4 hours in the first week and up to 8 hours after that period. Should any part of you feel uncomfortable, the participant should return immediately so that the appropriate adjustments are made in the slipper
  Interventions: Other: custom slippers with perforated synthetic leather cover.
- Control group (Sham Comparator): The control (sham) group volunteers will receive a pair of custom slippers with perforated synthetic leather cover as those used by GI.
  The difference will be that these slippers will not have the elements in the insoles.
  Interventions: Other: custom slippers with perforated synthetic leather cover.

INTERVENTIONS:
Other: custom slippers with perforated synthetic leather cover. — the intervention group volunteers will receive a pair of custom slippers with perforated synthetic leather cover.

SUMMARY:
Introduction: Persistent heel pain from plantar fasciitis and calcaneal spurs, as well as metatarsalgia, are very common and prevalent complaints in the Brazilian population. One of the recommended treatments for these conditions in the literature is the use of insoles. However, the use of this feature requires the individual to wear closed shoes and this is an obstacle to treatment in cities with hot weather. Thinking about an alternative treatment, the customized slippers with the corrective elements of the insoles can be an alternative to increase the adhesion to this type of treatment. Objective: To evaluate the effectiveness of the insoles adapted in slippers in the improvement of the pain and the function in individuals with persistent pains in the backfoot of the city of Santa Cruz, RN. Methodology: This is a double-blind, randomized, controlled clinical study in which 66 patients diagnosed with persistent back pain and metatarsalgias will be divided into two groups. The intervention group will receive a customized slipper with foot pieces and synthetic leather cover, and the control group will receive a slipper without customization, only with a synthetic leather cover as used by the intervention group. The evaluator and the patient will be considered blind. Evaluations will be performed at baseline (T0), after 12 weeks of wearing the slippers (T12) and a reassessment at week 16 (T16) for pain monitoring. The evaluation instruments used will be the EVA (visual pain scale) and the algometer in the painful region of the foot; FFI - Foot Function Index questionnaire and FAAM questionnaire - Foot and Ankle Ability Measure for functional evaluation, and finally the 6 - minute walking test for walking performance. Statistical analysis: Data will be analyzed by t-test, Mann-Whitney test, repeated-measures ANOVA and intention-to-treat analysis.

DETAILED DESCRIPTION:
The evaluations for the prescription of the insoles will be made at the Physiotherapy School Clinic of FACISA / UFRN and a podoscope will be used to evaluate the foot typology and other morphological aspects, a pen to print the feet and make a mold for making the insoles. insoles, and different prosthetic parts molded previously.

The volunteers will be invited to participate in the research and, upon accepting, will be informed of the research procedures, sign the informed consent form and only then will be evaluated by the blind evaluator of the study. It will also be informed that it can be drawn for any of the two groups (intervention group or control group). Allocation in groups will be done randomly, by lot.

All volunteers, regardless of groups, will be evaluated individually, in a comfortable room, barefoot and wearing shorts or shorts.

Evaluations will occur at the baseline (T0), after 12 weeks of use of the slippers (T12) and at the follow up 4 weeks after the end of the intervention (T16).

The following evaluation tools will be used:

* Pain by Visual Analog Scale and algometer;
* The function of the foot by the FFI (Foot Function Index) questionnaire;
* Foot and ankle functionality by FAAM (Foot and Ankle Ability Measure);
* Functional ability by the 6-minute walk test;
* After this step, the volunteers will be evaluated on the podoscope using the foot pieces for the postural evaluation (fig 3). In the protocol, the volunteer's posture will be evaluated using the foot pieces to verify their influence on static balance and postural asymmetries. The volunteers will be evaluated in the frontal and sagittal planes.
* Finally, the volunteers will carry out the plantations (fig 4) that will be sent to make the slippers.

6.2 Calculation of the sample The investigators will select 66 patients from the list of patients at the Physiotherapy School Clinic of the FACISA / UFRN, with diagnosis of calcaneal spurs, fasciitis and / or metatarsalgia, according to clinical evaluation criteria. The project will also be broadcast by local radio and media.

The sample size was calculated based on the EVA variable, considering a power of 90%, a significance of 5% and a loss rate of 10%. Based on the study by Chuter, Searle and Spink (2016), where with similar methods they found a difference of 1.3 points, considering the standard deviation of this variable being equal to 1.8. Based on these data, a sample of 66 subjects with 33 in each group was necessary to detect a clinically important difference. The calculation was based on comparisons of two samples by Gpower 3.1 software. The randomization will be through a computer program, and from this result, the chips will be placed in opaque and sealed envelopes to maintain allocation secrecy.

6.3 Inclusion criteria Patients of both sexes with a diagnosis of persistent back pain and / or pain in the head region of the metatarsals for more than 3 months, aged 18-60 years, accustomed to wearing slippers that are not performing other types of physical therapy and sign the ICF.

6.4 Exclusion Criteria Patients with foot wounds, previous foot and ankle surgeries, rheumatic diseases and / or skin diseases and those reporting that they can not wear slippers.

6.5 Interventions Intervention Group (GI) - the intervention group volunteers will receive a pair of custom slippers with perforated synthetic leather cover. They will be advised to wear the slipper for 4 hours in the first week and up to 8 hours after that period. Should any part disturb you, the participant should return immediately to the appropriate adjustments to be made in the slipper.

Control group (CG) - control group volunteers will receive custom slippers with the same coverage as those used by GI. The difference will be that these slippers will not have the elements podais, will be a slipper with smooth surface.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a diagnosis of persistent back pain and / or pain in the head region of the metatarsals for more than 3 months, aged 18-60 years, accustomed to wearing slippers that are not performing other types of physical therapy and sign the ICF.

Exclusion Criteria:

* Patients with foot wounds, previous foot and ankle surgeries, rheumatic diseases and / or skin diseases and those reporting that they can not wear slippers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change in VAS - Visual Analog Scale | in baseline and 12 week
  Visual Analog Scale - 0 - 10. Likert scale, 0 - no pain and 10 - worst pain

SECONDARY OUTCOMES:
Change in FFI - Foot Function Index questionnaire | baseline and 12 week
  Foot Function Index questionnaire - To obtain the total score for each domain, the following formula was applied: sum of the score obtained from all items answered by the patient / possible total score of the domain × 100 in order to obtain the percentage value. If the patient does not do any activity indicated by one of the items (for example, do not make use of auxiliary devices), this is considered as not applicable. Thus, the scoring of these items will not be considered in the total sum of the domain. The final percentage of all domains must be summed and divided by three (total number of domains) to obtain the final result of the questionnaire. Results may range from 0 to 100% and are directly proportional to limb functional impairment. The higher the percentage, the greater is the functional alteration presented by the patient
Change in FAAM - Foot and Ankle Ability Measure | baseline and 12 week
  The scores for each of the items are added together to obtain the item score total. The total number of items with a response is then multiplied by 4 to obtain the highest potential score. If all 21 items were answered, the highest potential score would be 84. If one item was unanswered the highest potential score would be 80, if two items were unanswered the total highest score would be 76, and so forth. The total item score is divided by the highest potential score and then multiplied by 100 to produce the FAAM score, which ranges from 0 to 100. The Sports subscale is scored in a similar manner; the highest potential score is 32. As with the ADL subscale, the item score total is divided by the highest potential score and multiplied by 100. A higher score represents a higher level of physical function for both the ADL and Sports subscales.
Change in 6MWT - 6-minute walk test | baseline and 12 week
  1. The course can vary from 20 to 50 meters away, depending on the size of the aisle.
  2. Marking a line transverse to the demarcated space for the displacement at the beginning of the test.
  3. If test repeats are required, for comparison or evaluation of the outcome, subsequent tests should be performed at the same time as the 1st test day.
  (d) If a test is to be performed at least 10 minutes blood pressure, heart rate, and O 2 saturation. e) At the end of the test, the evaluator must be informed that he / she should walk slowly across the direction of the test to measure the distance by the evaluator, which should also demonstrate the scale of perceived effort and question the intensity of the test. test.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cardoso de Souza, PT,PhD, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Marcelo Souza, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there is not a plan to make individual participant data (IPD) available to other researchers.